CLINICAL TRIAL: NCT04879706
Title: Proenkephalin A at Initiation and Discontinuation of Kidney Replacement Therapy
Brief Title: Proenkephalin A and Kidney Replacement Therapy
Status: Terminated | Type: Observational
Why Stopped: Poor patient enrollment
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: AZ 37/21
Record Dates: First submitted 2021-05-03; First posted 2021-05-10 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AKI necessitating KRT: Patients with AKI necessitating KRT
  Interventions: Other: None planned

INTERVENTIONS:
Other: None planned — No intervention planned

SUMMARY:
Acute kidney injury (AKI) is a common problem encountered in the intensive care unit (ICU), estimated to occur in up to 60% of all critically ill patients, depending on the definition. Recent large randomized clinical trials in critical care nephrology have focused on the optimal timing of initiation of acute kidney replacement therapy (KRT). However, less is known about the ideal circumstances in which KRT may be successfully discontinued.

The novel serum-biomarker proenkephalin A 119-159 (penkid) has been found to be strongly negatively correlated with measured GFR. Whether penkid may have a role in initiation and discontinuation of KRT remains unknown.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common problem encountered in the intensive care unit (ICU), estimated to occur in up to 60% of all critically ill patients, depending on the definition. Recent large randomized clinical trials in critical care nephrology have focused on the optimal timing of initiation of acute kidney replacement therapy (KRT). However, less is known about the ideal circumstances in which KRT may be successfully discontinued. KRT is a complex and expensive therapy, with complications including catheter-associated infections, hemorrhage, hemodynamic instability, and potential delayed renal recovery.

The novel serum-biomarker proenkephalin A 119-159 (penkid) is a stable fragment derived from the precursor enkephalins, which are known as small endogenous opioid peptides and are produced throughout the human body, including the kidneys. Plasma concentrations of penkid have been found to be strongly negatively correlated with measured glomerular filtration rate. Whether penkid may have a role in initiation and discontinuation of KRT remains unknown.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age with AKI requiring KRT

Exclusion Criteria:

* Chronic kidney disease with estimated glomerular filtration rate <30 mL/min/1.73 m2
* Non-end stage renal disease with extracorporeal ultrafiltration due to diuretic- resistant fluid overload
* Decision to limit therapeutic interventions
* History of solid-organ transplants
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with severe AKI necessitating KRT at the University Hospital Giessen, Giessen, Germany
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2023-01-21 (Actual)

PRIMARY OUTCOMES:
Penkid levels at KRT initiation | Up to 2 weeks
  Serial assessment of penkid in patients undergoing KRT
Penkid levels at discontinuation of KRT | Up to 2 weeks
  Serial assessment of penkid in patients undergoing KRT

CONTACTS AND LOCATIONS:
Overall Officials: Werner Seeger, MD, Study Director — University of Giessen
Locations (1):
- University Hospital Gießen and Marburg, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim H, Hur M, Struck J, Bergmann A, Di Somma S. Proenkephalin Predicts Organ Failure, Renal Replacement Therapy, and Mortality in Patients With Sepsis. Ann Lab Med. 2020 Nov;40(6):466-473. doi: 10.3343/alm.2020.40.6.466. Epub 2020 Jun 17. PMID 32539302